CLINICAL TRIAL: NCT05165394
Title: A Randomized, Double-Blind, Placebo-Controlled, Proof-of-Concept Study to Evaluate the Efficacy and Safety of Once-Weekly Oral NBI-1065846 in the Treatment of Anhedonia in Major Depressive Disorder (TERPSIS STUDY)
Brief Title: Study to Evaluate the Efficacy and Safety of Once-Weekly Oral NBI-1065846 in the Treatment of Anhedonia in MDD
Acronym: TERPSIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1065846-MDD2020
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Anhedonia; Major Depressive Disorder
Keywords: Anhedonia; Major Depressive Disorder; MDD; NBI-1065846; TERPSIS; Neurocrine; Antidepressant; Depression; TAK-041
MeSH Terms: conditions — Anhedonia; Depressive Disorder, Major; Depression | interventions — TAK-041

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participant follows Placebo schedule (57 days)
  Interventions: Drug: Placebo
- Antidepressant (Experimental): Participant follows NBI-1065846 schedule (57 days)
  Interventions: Drug: NBI-1065846

INTERVENTIONS:
Drug: Placebo — Tablets for oral administration
  Arms: Placebo
Drug: NBI-1065846 — Tablets for oral administration
  Other Names: TAK-041
  Arms: Antidepressant

SUMMARY:
To evaluate the efficacy of NBI-1065846 compared with placebo on improving symptoms of anhedonia in participants with major depressive disorder (MDD).

ELIGIBILITY:
Key Inclusion Criteria:

Participants must meet all of the following key inclusion criteria:

1. Completed written informed consent.
2. Aged 18 to 65 years, inclusive, at the time of informed consent.
3. Primary diagnosis of MDD.
4. Participants must meet one of the following criteria:

   * must have been taking ≥1 antidepressant medication(s) for ≥8 weeks prior to screening.
   * must have received ≥1 antidepressant medication(s) for ≥8 weeks in the current or most recent episode of depression.
5. Snaith Hamilton Pleasure Scale (SHAPS) score is ≥30 at screening and Day 1.

Key Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following key criteria:

1. Any psychiatric disorder disallowed per protocol and electroconvulsive therapy (ECT) within 6 months prior to screening. Comorbid anxiety disorders are not exclusionary.
2. Have a significant risk of suicidal or violent behavior.
3. A history of seizure disorder, stroke, Alzheimer disease, Parkinson disease, multiple sclerosis, head injury associated with loss of consciousness for more than 15 minutes, or other neurodegenerative disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (23):
- United States (22):
  - Neurocrine Clinical Site, Birmingham, Alabama
  - Neurocrine Clinical Site, Garden Grove, California
  - Neurocrine Clinical Site, Lemon Grove, California
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, Riverside, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, San Francisco, California
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, Pensacola, Florida
  - Neurocrine Clinical Site, Winter Park, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Skokie, Illinois
  - Neurocrine Clinical Site, Saint Charles, Missouri
  - Neurocrine Clinical Site, Raleigh, North Carolina
  - Neurocrine Clinical Site, Columbus, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Friendswood, Texas
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Murray, Utah
  - Neurocrine Clinical Site, Everett, Washington
- Neurocrine Clinical Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NBI-1065846: Participant follows NBI-1065846 schedule (57 days).
Period: Overall Study
Arm/Group | Placebo | NBI-1065846
Started | 47 | 46
Received at Least 1 Dose of Study Drug | 47 | 46
Completed | 41 | 42
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other Than Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NBI-1065846 | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.8) | 43.8 (14.0) | 43.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 40 | 37 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 3 | 2 | 5
  Race: Black or African American | 4 | 6 | 10
  Race: White | 36 | 35 | 71
  Race: Other | 1 | 1 | 2
  Race: Multiple | 2 | 2 | 4
Dimensional Anhedonia Rating Scale (DARS) Score [Mean (Standard Deviation); unit: units on a scale] — The DARS is a dynamic scale that measured desire, motivation, effort and consummatory pleasure across hedonic domains. The DARS is a self-report questionnaire that measured anhedonia across 4 domains: hobbies/past-times, food/drinks, social activities, and sensory experiences. The DARs was rated on a five-point Likert scale from 0 (not at all) to 4 (very much), higher values indicated less anhedonia. All items were summed up to a total score in the range of 0 to 68.
  units on a scale | 15.1 (10.5) | 18.7 (12.8) | 16.9 (11.8)
Total Montgomery Åsberg Depression Rating Scale (MADRS) Score [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a validated rating scale designed to measure changes in the severity of depressive symptoms. The MADRS consists of 10 items scored on a 7-point scale (0 to 6). Higher MADRS scores indicate more severe depression. The MADRS total score was calculated as the sum of the 10 individual item scores which ranged from 0 to 60.
  units on a scale | 30.8 (6.6) | 31.0 (5.5) | 30.9 (6.1)
Clinical Global Impression - Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The CGI-S scale, which is based on a 7-point scale (range: 1=normal, not at all ill, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, and 7 = extremely ill), was used to rate the severity of the participants illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  units on a scale | 4.7 (0.7) | 4.8 (0.6) | 4.8 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anhedonia Severity, as Measured by Change in DARS Score From Baseline to Day 57
Description: The DARS is a dynamic scale that measured desire, motivation, effort and consummatory pleasure across hedonic domains. The DARS is a self-report questionnaire that measured anhedonia across 4 domains: hobbies/past-times, food/drinks, social activities, and sensory experiences. The DARs was rated on a five-point Likert scale from 0 (not at all) to 4 (very much), higher values indicating less anhedonia. All items were summed up to a total score in the range of 0 to 68.
Time Frame: Baseline, Day 57
Population: Full Analysis Set (FAS): All randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for specified outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | NBI-1065846
Number analyzed (Participants) | 44 | 45
units on a scale | 17.4 (3.7) | 13.5 (3.6)
Statistical Analysis 1: Comparison: Placebo vs NBI-1065846; Test type: Superiority; p = 0.8663, ANCOVA — Significance level = 0.1; Least-Squares Mean Treatment Difference = -3.9, 90% CI 1-sided [lower limit -8.4], Standard Error of Mean 3.5 — Confidence interval and p-value are one-sided for test of null hypothesis that the LS mean difference between NBI-1065846 and placebo in DARS total score at Day 57 is greater than or equal to zero

2. Secondary Outcome: Change in Total MADRS Score From Baseline to Day 57 in Participants With Moderate or Higher Severity Depression
Description: The MADRS is a validated rating scale designed to measure changes in the severity of depressive symptoms. The MADRS consists of 10 items scored on a 7-point scale (0 to 6). Higher MADRS scores indicate more severe depression. The MADRS total score was calculated as the sum of the 10 individual item scores which ranges from 0 to 60.
Time Frame: Baseline, Day 57
Population: FAS: All randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for specified outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | NBI-1065846
Number analyzed (Participants) | 31 | 33
units on a scale | -13.9 (3.4) | -15.1 (3.0)
Statistical Analysis 1: Comparison: Placebo vs NBI-1065846; Test type: Superiority; p = 0.7008, ANCOVA; Least-Squares Mean Treatment Difference = -1.1, 95% CI 2-sided [-7.1 to 4.8], Standard Error of Mean 3.0 — NBI-1065846 - Placebo

3. Secondary Outcome: CGI-S Scores
Description: The CGI-S scale, which is based on a 7-point scale (range: 1=normal, not at all ill, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, and 7 = extremely ill), was used to rate the severity of the participants illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Time Frame: Baseline and Day 57
Population: FAS: All randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for specified outcome measure. Number analyzed = number of participants with evaluable data at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NBI-1065846
Number analyzed (Participants) | 46 | 45
Participants
  Baseline: Normal, not at all ill (1): number analyzed (Participants) | 46 | 42
  Baseline: Normal, not at all ill (1) | 0 | 0
  Baseline: Borderline ill (2): number analyzed (Participants) | 46 | 42
  Baseline: Borderline ill (2) | 0 | 0
  Baseline: Mildly ill (3): number analyzed (Participants) | 46 | 42
  Baseline: Mildly ill (3) | 1 | 1
  Baseline: Moderately ill (4): number analyzed (Participants) | 46 | 42
  Baseline: Moderately ill (4) | 16 | 11
  Baseline: Markedly ill (5): number analyzed (Participants) | 46 | 42
  Baseline: Markedly ill (5) | 23 | 26
  Baseline: Severely ill (6): number analyzed (Participants) | 46 | 42
  Baseline: Severely ill (6) | 6 | 4
  Baseline: Extremely ill (7): number analyzed (Participants) | 46 | 42
  Baseline: Extremely ill (7) | 0 | 0
  Day 57: Normal, not at all ill (1): number analyzed (Participants) | 44 | 45
  Day 57: Normal, not at all ill (1) | 6 | 7
  Day 57: Borderline ill (2): number analyzed (Participants) | 44 | 45
  Day 57: Borderline ill (2) | 7 | 7
  Day 57: Mildly ill (3): number analyzed (Participants) | 44 | 45
  Day 57: Mildly ill (3) | 12 | 11
  Day 57: Moderately ill (4): number analyzed (Participants) | 44 | 45
  Day 57: Moderately ill (4) | 10 | 12
  Day 57: Markedly ill (5): number analyzed (Participants) | 44 | 45
  Day 57: Markedly ill (5) | 9 | 7
  Day 57: Severely ill (6): number analyzed (Participants) | 44 | 45
  Day 57: Severely ill (6) | 0 | 1
  Day 57: Extremely ill (7): number analyzed (Participants) | 44 | 45
  Day 57: Extremely ill (7) | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs NBI-1065846; CGI-S scores at Day 57 for NBI-1065846 compared to placebo; Test type: Superiority; p = 0.9051, Cochran-Mantel-Haenszel Chi-square test

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Day 106
Description: Safety Analysis Set: All randomized participants who took at least 1 dose of study treatment.
  Participants were analyzed according to their randomized treatment group, unless they received the incorrect study treatment for the entire treatment duration.
  Time frame includes treatment period (Days 1 to 57) and safety follow-up period (up to Day 106).
Arm/Group | Placebo | NBI-1065846
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/46
Other Adverse Events (participants affected / at risk) | 4/47 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | NBI-1065846 (N=46)
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | NBI-1065846 (N=46)
Headache (Nervous system disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT05165394/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT05165394/SAP_001.pdf